CLINICAL TRIAL: NCT05158530
Title: Effect Of Exercise Training In Patients With Lung Cancer During Chemotherapy Treatment
Brief Title: Effect of Exercise Training in Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01093 Muheebur Rehman
Record Dates: First submitted 2021-12-13; First posted 2021-12-15 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Lung Cancer, Nonsmall Cell
Keywords: Nonsmall Cell Lung cancer, Chemotherapy, Exercise training
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group (Experimental): Pulmonary exercises + Aerobic training, 40%-60% intensity 3 days/ week for 4 weeks
  Interventions: Other: Aerobic training
- Control group (Placebo Comparator): Pulmonary exercises, 3 sessions per week and 3-5 repetitions in a session for 4 weeks.
  Interventions: Other: Pulmonary Exercises

INTERVENTIONS:
Other: Aerobic training — Aerobic training ( with cycle ergometer, 5-minute warm-up 15 - 30 minute cycle +5 minute cooldown) 40%-60% intensity calculated through Karvonen formula 3 days/ week
  Arms: Interventional Group
Other: Pulmonary Exercises — 4 weeks protocol
  1. Deep breathing Exercises* 10 Reps 3 sets
  2. Postural drainage (10 minutes * 2 sets /day)
  3. Incentive spirometry* 10 Reps 3 sets
  4. Bed activities (Active ankle and hand pumping exercise * 10 Reps 3 sets)
  Arms: Control group

SUMMARY:
To determine the effects of exercise training in patients with lung cancer during chemotherapy treatment. In currently accessible literature, majority studies, met-analysis, and systemic reviews are related to surgical procedures and post-op pulmonary Rehabilitation of patients with Lung cancer. In literature, Gap related to the control group was observed also. The current study aimed to fulfill this gap by planning a structured intervention plan for the control group as well. It will also add in literature the deficiency of oncology rehab for patients receiving chemotherapy only.

DETAILED DESCRIPTION:
Literature suggested that a pulmonary rehabilitation program for patients with non-small cell lung cancer undergoing induction chemo-radiotherapy seems to improve respiratory function. It is particularly recommended for smokers and patients with respiratory impairment.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosed patients of stage 1 and 2 Non-small cell lung carcinoma (NSCLC) including Adenocarcinoma & squamous cell carcinoma The diagnosis was established within 6 wk prior to enrollment and was confirmed by histology.

Participants are undergoing lung cancer chemotherapy Participant has the willingness to participate in training WHO physical fitness scores 0-1 Able to perform 6-minute walk test (6MWT) at baseline

Exclusion Criteria:

* • Participant with history of trauma and surgery

  * Patients with lung disease other than lung cancer
  * Uncontrolled hypertension or unstable coronary artery disease.
  * Severe OA, bone or CNS metastases.
  * hemoglobin <10 g/dL
  * Lower than 3,500 white blood cells per microliter of blood

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
6 min walk test: Distance (meters) | 4 weeks
  Changes from the baseline, 6 min walk test (6 MWT) was used to measure Functional capacity. It is a sub maximal exercise test which can aid in assessing functional capacity of patients with cardiopulmonary diseases, in this test we find out the maximum distance in meters which an individual covers in 6 min without any support.
Forced Expiratory Volume in 1 second (FEV1) | 4 weeks
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze Forced Expiratory Volume in 1 second FEV1 in Liters
Forced vital Capacity (FVC) | 4 weeks
  Changes From the Baseline, the digital spirometer is used in clinical setting to analyze Forced vital Capacity in Liters
Rate of perceived exertion (RPE) | 4 weeks
  Changes From the Baseline, measured through Borg RPE scale which measures a person's perception of their effort and exertion breathlessness, and fatigue during physical work rating between 1 and 10. The higher the number, the more intense the exercise. An RPE of 1 is often referred to as just above rest, hardly any exertion, while an RPE of 10 is a maximal effort.

SECONDARY OUTCOMES:
Mindfulness | 4 weeks
  Changes From the Baseline, measured through MAAS. The MAAS is a 15-item scale designed to assess a core characteristic of dispositional mindfulness, namely, open or receptive awareness of and attention to what is taking place in the present. The scale shows strong psychometric properties and has been validated with college, community, and cancer patient samples.Higher scores reflect higher levels of dispositional mindfulness
Hospital Anxiety and Depression | 4 weeks
  The Hospital Anxiety and Depression Scale (HADS) is a frequently used self-rating scale developed to assess psychological distress in non-psychiatric patients. HADS is a fourteen-item scale with seven items each for anxiety and depression subscales. Scoring for each item ranges from zero to three. A subscale score >8 denotes anxiety or depression

CONTACTS AND LOCATIONS:
Overall Officials: Mehwish Waseem, MSPT(CPPT), Principal Investigator — Riphah International University
Locations (1):
- Institute of Radiotherapy and Nuclear Medicine, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davis KM, Kelly SP, Luta G, Tomko C, Miller AB, Taylor KL. The association of long-term treatment-related side effects with cancer-specific and general quality of life among prostate cancer survivors. Urology. 2014 Aug;84(2):300-6. doi: 10.1016/j.urology.2014.04.036. Epub 2014 Jun 26. PMID 24975711
- [Background] Vainshelboim B, Fox BD, Saute M, Sagie A, Yehoshua L, Fuks L, Schneer S, Kramer MR. Limitations in exercise and functional capacity in long-term postpneumonectomy patients. J Cardiopulm Rehabil Prev. 2015 Jan-Feb;35(1):56-64. doi: 10.1097/HCR.0000000000000085. PMID 25350720